CLINICAL TRIAL: NCT01574521
Title: A Fetal Seroepidemiologic Study in Hepatitis B Virus Transmitted Via Male Germ Line
Brief Title: Seroepidemiologic Study of Spermatozoal Transmission of Hepatitis B Virus (HBV)
Status: Completed | Type: Observational
Sponsor: YiYang Zhu (Other)
Responsible Party: Sponsor-Investigator, YiYang Zhu, Center for Prenatal Diagnosis, Taizhou Hospital
Organization: Taizhou Hospital (Other)
Other Study IDs: tz2008032
Record Dates: First submitted 2012-04-08; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum,amniotic fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Only father carrier: fetuses whose fathers were HBV carriers whereas mothers negatively.
- only mother carrier: fetuses whose mothers were HBV carriers whereas fathers negatively.
- both parents carriers: fetuses whose both parents were HBV carriers

SUMMARY:
Animal experiments demonstrated that father might transmit HBV vertically via male germ line, however, whether it is really existed in human remains to be determined. Since HBV is a blood-borne virus, the unvaccinated pregnant women would be at risk for HBV exposure if their fetuses carried the virus from fathers. If women had been vaccinated for HBV before conception, what would happen to a maternal immune system if her fetus carried HBV from spermatozoa? However, the literature on transmission of HBV by spermatozoa in vivo is rare, the viral replicating status and fetal immune response in uterus are unknown. The aim of study was to detect father-to-fetus transmission of hepatitis B virus (HBV) in uterus.

DETAILED DESCRIPTION:
Transmission of hepatitis B virus (HBV) from mother-to-infant is the predominant route in most high prevalence areas such as China. However, father-to-child transmission also plays another important role in the prevalence of hepatitis B. Children infected with HBV from their carrier fathers would be horizontally by postnatal intimate contact or vertically via male germ line. The latter is considered an intrauterine infection, however, whether it is really existed in human remains to be determined.

In past decades, several experiments reported there presences of integrated HBV DNA in human spermatozoal chromosomes. Studies on embryos hybridized with mammalian ova and human spermatozoa were also confirmed that sperm-integrated HBV DNA can replicate and express the HBV protein in two-cell' hybrid embryos. All above findings demonstrated that father might transmit HBV to fetus by spermatozoa in theory.

Since HBV is a blood-borne virus, the unvaccinated pregnant women would be at risk for HBV exposure if their fetuses carried the virus from fathers. On other hand, maternal antibodies can pass through the placenta and enter the fetal circulation freely. If women had been vaccinated for HBV before conception, thus some attractive questions are raised that what would happen to a maternal immune system if her fetus carried HBV from spermatozoa? Would the fetus be passive immunized by hepatitis B immunoglobulin leaked from maternal circulation? However, the literature on transmission of HBV by spermatozoa in vivo is rare, the viral replicating status and fetal immune response in uterus are unknown. Only one study had detected HBV DNA and serological makers on eight aborted fetuses suspected with HBV transmission via spermatozoa, but it is a small sample study and the maternal serological status is uncertain.

Specimens applied for evaluating intrauterine infection include amniotic fluids, placental tissue and neonatal peripheral blood. Because postnatal sample is inevitably to be contaminated by maternal blood during delivery, it would be useless to determine the time when the infection was occurred (before or during the partum). A better alternative is detecting fetal infection before the partum by prenatal diagnostic technique. Comparing to the postnatal specimens, intrauterine specimens obtained from amniocentesis or cordocentesis can minimize the contamination of maternal blood. It is also a safety technique and the risk of nosocomial infection caused by invasive procedures is very low. The aim of this study was to investigate the fetal hepatitis B seroepidemiology by prenatal diagnostic technique and to find the evidence of HBV vertical transmission via spermatozoa.

ELIGIBILITY:
Inclusion Criteria:

* one or both of pregnant Woman and her husband were HBV carriers
* indicated for amniocentesis or cordocentesis

Exclusion Criteria:

* indicated for chorionic villous sampling

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The research consisted of the pregnant women who visited for prenatal diagnosis during the January 2008 and June 2010.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
positive rate of HBV in uterus | one year
  HBV infection confirmed by serological makers(HBsAg, HBeAg, anti-HBs, anti-HBe anti-HBc)and HBVDNA. Samples were assessed by enzyme immunoassays and FQ-PCR

SECONDARY OUTCOMES:
response rate of postnatal vaccination | half a year after immunization series
  neonates received three doses of recombinant vaccines were given on a 0-, 1-, and 6-month schedule, and other 100 IU of HBIG was administrated within 24 hours after birth. Post-vaccination testing for efficacy evaluation was performed at one-year old (half a year after immunization series).

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Yang Zhu, MD, Study Director — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Locations (1):
- Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang, China